CLINICAL TRIAL: NCT02284945
Title: A Randomized Controlled Trial Comparing Open Spinal Stabilisation and Percutaneous Solution (TPS) Surgery in Patients With Metastatic Spinal Disease.
Brief Title: Randomized Controlled Trial of Open Stabilisation Versus TPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NE11/9972; 11/YH/0404 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-10-28; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Metastatic Spinal Disease
MeSH Terms: conditions — Spinal Diseases

ARMS (2):
- Posterior percutaneous instrumentations (Experimental)
  Interventions: Procedure: Keyhole surgery
- Traditional open surgery with pedicle screw fixation (Other)
  Interventions: Procedure: Open fixation

INTERVENTIONS:
Procedure: Open fixation
  Arms: Traditional open surgery with pedicle screw fixation
Procedure: Keyhole surgery
  Arms: Posterior percutaneous instrumentations

SUMMARY:
Spread of cancer to the spinal column is a growing problem in patients with cancer. It can cause a number of problems including pain, instability and neurologic problems. If left untreated, progressive weakness, numbness and bladder/bowel disturbance occurs. The aim of treatment is to help with pain and to reduce the risk of these neurological problems. This treatment has traditionally been radiotherapy to the spine. Surgery has always meant large open operations with a long recovery time and significant risk of complications. There has been new technology that has allowed less invasive operations to take place to stabilise the spine. The aim is to relieve the pressure on the spinal cord in addition to stabilising the spinal cord. These techniques are called 'minimally invasive' and include surgical techniques such as cement augmentation and percutaneous instrumentation.

The aim of this study is to compare traditional open operations with these new minimally invasive techniques to see if they do result in reduced complications and quicker recovery in addition to achieving the goals of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has an age ≥ 18 years
* Is suitable for radiotherapy
* Has been assessed by the oncologist
* Has symptoms of pain
* Is diagnosed with metastatic spinal pain from MRI findings with or without biopsy
* Technically possible to perform the surgery
* Is willing and able to comply with required followup questionnaires
* Is able to understand the risks and benefits of participating in the study
* Understands and has signed the informed consent form.
* Life expectancy of > 3 months

Exclusion Criteria:

* Active systemic infection or infection localized to the site of implantation
* Allergy or sensitivity to Polyether ether ketone (PEEK), Titanium or Tantalum
* A bleeding disorder precluding from invasive surgery
* Rapid neurological deterioration requiring urgent surgery which would be delayed to the detriment of the patient by including in this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain (VAS) scores | 3 months
Visual analogue pain (VAS) scores | 6 months
Visual analogue pain (VAS) scores | 1 year
Visual analogue pain (VAS) scores | 2 years
Oswestry disability score | 3 months
Oswestry disability score | 6 months
Oswestry disability score | 1 year
Oswestry disability score | 2 years
EuroQoL Questioonaire (EQ-5D) | 3 months
EuroQoL Questioonaire (EQ-5D) | 6 months
EuroQoL Questioonaire (EQ-5D) | 1 year
EuroQoL Questioonaire (EQ-5D) | 2 years